CLINICAL TRIAL: NCT07138820
Title: 18F-choline-PET-CT vs Ultrasonography and 99-technetium Sestamibi Scintigraphy in Preoperative Localization for pHPT - A Randomized Trial
Brief Title: 18F-choline Positron-emission-tomography - Computed-tomography Compared to Conventional Imaging for Localizing Diseased Parathyroid Glands in Primary Hyperparathyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Martin Almquist, Associate professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18FCHPET_PHPT
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Primary Hyperparathyroidism
Keywords: surgery; positron emission tomography; scintigraphy; ultrasonography; primary hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Parathyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18-F-choline-PET (Experimental): Investigation with 18-F-choline-PET-CT
  Interventions: Procedure: Parathyroidectomy
- Conventional (Active Comparator): Conventional (standard) imaging with ultrasonography and sestamibi scintigraphy
  Interventions: Procedure: Parathyroidectomy

INTERVENTIONS:
Procedure: Parathyroidectomy — Imaging with 18-F-choline-PET-CT

SUMMARY:
The goal of this open, single-center, prospective, randomized, clinical study is to compare imaging with [18F]fluoromethyl-dimethyl-2-hydroxyethylammonium (18F-choline) positron-emission-tomography - computed-tomography, 18F-ch-PETCT, to conventional imaging with ultrasonography and sestamibi scintigraphy in localizing diseased parathyroid glands in patients diagnosed with primary hyperparathyroidism, pHPT. The question this study aims to answer is: can 18-F-ch-PET-CT more precisely localize diseased parathyroid glands in patients with pHPT before surgery? The objective of the study is to help improve precision in parathyroid surgery, thereby increasing cure rates, minimizing complications, and shortening operation times.

DETAILED DESCRIPTION:
1 Improving precision in parathyroid surgery 18F-choline-PET-CT vs ultrasonography and 99-technetium sestamibi scintigraphy in preoperative localization for pHPT - A randomized trial Martin Almquist, 2022-03-08 Purpose and aims The purpose of the present open, single-center, prospective, randomized, clinical study is to investigate whether precision imaging with [18F]fluoromethyl-dimethyl-2-hydroxyethylammonium (18F-choline) positron-emission-tomography - computed-tomography, 18F-ch-PETCT, is superior to conventional imaging in localizing diseased parathyroid glands in primary hyperparathyroidism, pHPT. Our overall objective is to improve precision in parathyroid surgery, increase cure rates, minimize complications and shorten operation times. State-of-the-art Primary hyperparathyroidism (pHPT) is a common endocrine disorder, causing kidney stones, renal insufficiency, and osteoporosis, which increases the risk of fractures, especially hip fractures, which carry a substantial mortality risk (1). PHPT is caused by increased production of parathyroid hormone (PTH) in one or several enlarged parathyroid glands. Surgical removal of the pathologic gland(s) cures the disease (2). Successful preoperative localization of such glands limits the surgical dissection, increases the cure rate, minimizes complications, and decreases operation time (3). However, there is no perfect imaging method, which in all patients correctly identifies each and every pathologic gland (4). Commonly used imaging methods are neck ultrasonography and 99-technetium sestamibi scintigraphy (5). In patients with inconclusive imaging, multiphase four-dimensional computed tomography, 4DCT, can further help localize diseased parathyroids (6). The rate of inconclusive or negative studies is high (5). The current first-line imaging strategy with ultrasound and scintigraphy causes up to a half of patients to undergo no less than three localization procedures, adding to costs and inconvenience for patients. Replacing the current strategy with one modality might thus be beneficial for patients and cost-effective for the health care system. Imaging with [18F]fluoromethyl-dimethyl-2-hydroxyethyl-ammonium- PET-CT, 18F-ch-PET-CT, previously used for detection and staging in prostate cancer, might more precisely localize parathyroid glands than ultrasound and scintigraphy (7). However, 18F-ch-PET-CT is also more expensive than ultrasound and sestamibi scintigraphy, and not available at all centers. Hence, 18F-ch-PET-CT has mostly been used as a second-line method, for instance in patients with inconclusive ultrasound and/or scintigraphy, or in patients with persistent disease after previous parathyroid surgery (7). Significance and scientific novelty 18F-choline-PET-CT has not been used as the first-line modality in localizing parathyroid glands, and there has been no randomized trial comparing its efficacy to conventional imaging in this setting. A randomized trial would yield solid evidence and its results would be both novel and clinically important. 2 Preliminary and previous results Between 1st January 2017 and 31st December 2020, a total of 241 patients with first-time, nonhereditary pHPT were operated on at the Department of Surgery at Skåne University Hospital, Lund. Out of these, 225 patients (93 %) underwent ultrasonography, and 223 patients (92 %) underwent 99-technetium sestamibi scintigraphy. Ultrasound was inconclusive in 39 % of 225 patients, and sestamibi scintigraphy was inconclusive in 47 % of 223 patients. Hence, 116 patients (48 % of all patients) also underwent 4DCT. 4DCT was inconclusive in 28 % of patients.

Thus, a total of 42 (17 % of all patients) had inconclusive results in all three investigations. In patients with localized disease, the cure rate was 95 %; in patients where all three examinations were inconclusive, the cure rate was only 81 %. Thus, precision in preoperative localization is needed. At the Department of Clinical Physiology and Nuclear Medicine, Skåne University Hospital, 18Fch- PET-CT has been used in 5,500 patients between 2008 and 2019 for imaging of prostate cancer. No adverse reactions were reported. An on-site cyclotron, PETtrace 880, GE Healthcare, is used to produce the radiotracer [18F]fluoromethyl-dimethyl-2-hydroxyethylammonium.

Project description Theory and methods This is a non-blinded, single-center, prospective, randomized, clinical study comparing 18F-ch- PET-CT to 99-technetium sestamibi scintigraphy and ultrasonography for localizing parathyroid glands in primary hyperparathyroidism. Inclusion and exclusion criteria Adult patients with primary hyperparathyroidism referred to the Department of Surgery at Skåne University Hospital, Lund, deemed candidates for surgery by the attending surgeon, using criteria specified in clinical national and international guidelines, patient preferences, and surgeon judgment of indication and operability, are invited to participate. Invited patients are given oral and written information. After signed informed consent, patients are randomized to either 18F-ch-PET-CT or ultrasound and scintigraphy. Allocation is open, since blinding is not possible, neither for providers nor for patients. Patients with previous parathyroid or thyroid surgery, or with the need for concurrent thyroid surgery, or with lithium therapy, hereditary parathyroid disease, such as multiple endocrine neoplasia type 1, MEN1, or with severe renal insufficiency, are not eligible. Outcomes Since cure rates are high, even after negative imaging, 18F-ch-PET-CT might only increase cure rates slightly. However, more precise preoperative localization with 18F-ch-PET-CT should decrease operation time, facilitating surgical planning, with similar or higher cure rates than conventional imaging with ultrasound, scintigraphy, and (in half of the patients) 4DCT.

The primary outcome, therefore, is operation time, measured from incision to the last suture.

Secondary outcomes are cure rates, defined as normocalcemia without treatment with calcium or vitamin D at first follow-up, one month postoperatively; rates of complications such as damage to the recurrent laryngeal nerve and hypocalcemia; rates of persistent disease, i.e.

hypercalcemia at one month postoperatively; sensitivity, specificity, positive and negative 3 predictive values, per-lesion and per-patient; the total amount of irradiation; and total imaging and procedure costs. Safety Patients randomized to the conventional arm are not at increased risk due to the study. Patients randomized to 18F-ch-PET-CT are at risk for side-effects of this investigation. Potential side effects include adverse reactions to the radionuclide 18F-choline, radiation, and incidental findings. The mean effective dose of radiolabelled choline PET, ranging from 2.5 to 3.8 milliSievert, mSV, was lower than that of parathyroid scintigraphy performed with different techniques in the metaanalysis by Treglia et al. The addition of low-dose CT imaging for the hybrid approach yielded minimal further radiation exposure, 0.8 mSv (7). Thus, patients randomized to 18F-ch-PET-CT will not be subjected to more irradiation than the patients in the conventional arm.

Adverse reactions to [18F]fluoromethyl-dimethyl-2-hydroxyethyl-ammonium (18F-choline) are rare; none were reported in a meta-analysis on 18F-ch-PET-CT for prostate cancer, and none have been reported at the Department of Nuclear Medicine, Skåne Lund University Hospital, in a series of 5,500 patients. Power Currently, patients with pHPT have a mean (SD) operation time of 45 (25) minutes, whereas those with well-localized disease have currently a mean (SD) operation time of 31 (15) minutes.

To show a difference of 45 vs 30 minutes or greater, with alpha set to 0.05 and 80 % power, 44 patients in each arm are needed (8). To account for attrition, an extra 6 patients in each arm will be included. Thus, the trial will need to include and randomize 100 patients, 50 to each arm.

Feasibility and time plan During the last 3 years, a mean of 80 patients annually fulfilling inclusion criteria were operated on at the Department of Surgery at Skåne University, Lund. Assuming an inclusion rate of 85 %, inclusion would take 18 months. Given current wait times for surgery at the department, all patients would be expected to be operated on within 24 months. We will be able to analyze their outcomes within two and half years. A report of the study should be expected within 3 years.

Project organization Logistics Referrals to the surgical department are checked daily by one of the attending surgeons.

Referrals on patients deemed candidates for this study will be marked, and the research nurse will send patients a letter informing them about the study, and answer relevant questions by phone. Patients potentially eligible for the study will be seen by the PI. Patients' inclusion and exclusion criteria will be checked and noted, and eligible patients will be invited to participate. It is estimated that the PI will use 10 % of working time to oversee the study, inform and randomize patients. The research nurse will use 10 % of working time to further inform patients and managing referrals and appointments for imaging. Two specialist nuclear medicine physicians will devote 5 % of their time to management of the study, more specifically for image interpretation. 4 Data collection All data for the study will be collected using the Scandinavian Quality Register of Thyroid and Parathyroid Surgery, SQRTPA (9). This quality register is recognized by the Swedish Association of Local Authorities and Regions, the National Board of Health and Welfare, the Swedish Surgical Society, and the Swedish Association for Otorhinolaryngology and Head and Neck Surgery. The SQRTPA is managed by AddPro AB (10), a specialized IT-consulting company based in Lund, Sweden. All data are securely stored on servers located in Sweden.

The PI will have full access to the study data. Randomization Patients will be randomized using the built-in function of the SQRTPA (9). Data analysis and statistics With an expected difference of 45 (SD:25) and 30 minutes in the experimental and conventional arm, and alpha 0.05, beta 0.80, a total of 44+44 patients are needed (8). To account for attrition, 100 patients will be included. Primary and secondary outcomes will be analyzed using the intention-to-treat model, where patients are compared according to the group they were randomized to. We will also conduct multivariable regression models to identify factors associated with high and low specificity and sensitivity of 18F-ch-PET-CT, to further understand potential strengths and weaknesses with the method. Equipment No special equipment will be needed. Need for research infrastructure. This study will not need any extraneous research infrastructure. International and national collaboration This is a single-center study. No national or international collaboration will be sought for this study. Other applications or grants. Local grants will be sought after ethical approval (Skåne University Hospital Funds, Funds of the Southern Health Care Region, ALF) Independent line of research. This an independent line of research. The PI has no relations with other researchers or projects that will affect the present study. Clinical significance. Currently, a precise method to localize the parathyroid glands preoperatively is lacking.

Precision imaging with 18F-ch-PET-CT has the potential to reduce the number of investigations necessary to localize and identify the diseased gland and will decrease operation time, with maintained or improved cure rates, lower hospital stay, and lower costs. If successful, this precision imaging modality will be immediately implemented into the clinical routine at the Departments of Surgery and Nuclear Medicine in Lund; likely, other hospitals in Sweden and internationally will follow. 5 References

1. Kristensen PK, Perez-Vicente R, Leckie G, Johnsen SP, Merlo J. Disentangling the contribution of hospitals and municipalities for understanding patient level differences in oneyear mortality risk after hip-fracture: A cross-classified multilevel analysis in Sweden. PLoS One.

   2020;15(6):e0234041.
2. Wilhelm SM, Wang TS, Ruan DT, Lee JA, Asa SL, Duh QY, et al. The American Association of Endocrine Surgeons Guidelines for Definitive Management of Primary Hyperparathyroidism. JAMA Surg. 2016;151(10):959-68.
3. Bergenfelz A, van Slycke S, Makay O, Brunaud L. European multicentre study on outcome of surgery for sporadic primary hyperparathyroidism. Br J Surg. 2020.
4. Bunch PM, Kelly HR. Preoperative Imaging Techniques in Primary Hyperparathyroidism:

A Review. JAMA Otolaryngol Head Neck Surg. 2018;144(10):929-37. 5. Kunstman JW, Kirsch JD, Mahajan A, Udelsman R. Clinical review: Parathyroid localization and implications for clinical management. J Clin Endocrinol Metab. 2013;98(3):902- 12. 6. Kluijfhout WP, Pasternak JD, Beninato T, Drake FT, Gosnell JE, Shen WT, et al.

Diagnostic performance of computed tomography for parathyroid adenoma localization; a systematic review and meta-analysis. Eur J Radiol. 2017;88:117-28. 7. Treglia G, Piccardo A, Imperiale A, Strobel K, Kaufmann PA, Prior JO, et al. Diagnostic performance of choline PET for detection of hyperfunctioning parathyroid glands in hyperparathyroidism: a systematic review and meta-analysis. Eur J Nucl Med Mol Imaging.

2019;46(3):751-65. 8. https://clincalc.com/stats/samplesize.aspx. 9. https://sqrtpa.se 10. www.addpro.se

ELIGIBILITY:
Inclusion Criteria:

Proven primary hyperparathyroidism Indication for surgery Adult (>18 years)

Exclusion Criteria:

Inability to give informed consent Allergy to contrast Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Operation time | During surgery
  Operation time in minutes, skin-to-skin

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
Personal integrity.